CLINICAL TRIAL: NCT01629940
Title: Phenotypic and Genetic Properties in Males at Risk for X-linked Hypohidrotic Ectodermal Dysplasia: Evaluation of an Early Diagnosis Technology and Tests to Assess Nutritional Status
Acronym: ECP-013
Status: Completed | Type: Observational
Sponsor: Edimer Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ECP-013
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: X-linked Hypohidrotic Ectodermal Dysplasia; Hypohidrotic Ectodermal Dysplasia
Keywords: X-linked Hypohidrotic Ectodermal Dysplasia; Hypohidrotic Ectodermal Dysplasia; XLHED; HED
MeSH Terms: conditions — Ectodermal Dysplasia 1, Anhidrotic

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Male HED-Affected Individuals: Male subjects affected by HED
- Male controls: Male subjects not affected by HED

SUMMARY:
The investigators propose to obtain facial photographs for use in testing a computer algorithm that recognizes males at high risk for Hypohidrotic Ectodermal Dysplasia (XLHED). FDNA (www.fdna.com), a software company with expertise in the area of facial recognition, is collaborating with the Sponsor in algorithm development based on 2D photographs not requiring special photographic technologies. A frontal facial photograph will be taken at the time of study conduct. The anonymized photographs will be transmitted to FDNA for analysis. A limited number of unaffected controls will be also be recruited.

A subset of affected males between ages 5 and 25 years will have the option of having a blood draw for a set of laboratory studies assessing nutritional status.

DETAILED DESCRIPTION:
As the first exploratory objective for this study, we propose to obtain facial photographs for use in testing a computer algorithm that recognizes males at high risk for XLHED. While 3D facial profiling has been reported in HED, the technology does not meet the ease-of-use criteria for a universal screening tool. FDNA (www.fdna.com), a software company with expertise in the area of facial recognition, is collaborating with the Sponsor in algorithm development based on 2D photographs not requiring special photographic technologies. All males at risk for a diagnosis of XLHED and attending the 2012 NFED Family Conference will be eligible to participate. A short medical questionnaire will verify the clinical presentation, they will be requested to provide a baby photograph taken at up to 1 month of age (to be returned at study completion), and a frontal facial photograph will be taken at the time of study conduct. The anonymized photographs will be transmitted to FDNA for analysis. A limited number of unaffected controls will be recruited at the 2012 NFED Family Conference for the photography study, in addition to the control data already available in the FDNA database.

As a second exploratory objective, a subset of affected males between ages 5 and 25 years will have the option of having a blood draw for a set of laboratory studies assessing nutritional status. HED-affected patients in general (including XLHED) are reported to have evidence of growth restriction (weight for height) in this age range without clear mechanistic evidence. A screening panel of nutritional laboratory tests has been designed in collaboration with experts in the field at the University of California, San Francisco (UCSF). Anonymized samples will be analyzed at UCSF.

ELIGIBILITY:
Inclusion Criteria:

1. Males of any age who are registered and attending the 2012 NFED Family Conference;
2. Conform to one of the following requirements for providing informed consent/assent:

   * if more than 18 years of age, subjects must provide signed informed consent;
   * if less than 18 years of age and it is determined that the subject is capable of providing assent, both the assent of the subject and consent of the parent(s) or guardian of that subject must be granted. Under this condition, both parents of the subject should give their permission, unless 1 parent is deceased, unknown, incompetent, or not available;
   * if the subject is incapable of providing assent, the consent of the parent(s) or guardian of the subject must be granted. Under this condition, both parents should give their consent, unless 1 parent is deceased, unknown, incompetent, or not available.
3. As described in Section 3.2 above, subjects must meet one of the following criteria:

   * Male subjects of original gender with genetic confirmation of an EDA mutation or with the clinical characteristics of HED including a history of decreased sweating;
   * Unaffected, healthy male controls.

Exclusion Criteria:

1. Subjects who are not able or are not willing to comply with the procedures of this protocol.
2. Subjects with any major medical problem that will prevent them from participating in this study.
3. HED-affected male subjects who have had prior genetic testing confirming they do not have the X-linked form of the disorder.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study is being conducted among family members attending the 2012 National Foundation for Ectodermal Dysplasia (NFED) Family Conference, July 19-21, 2012, in Orlando, FL.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2012-06; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Exploratory Objective - To collect demographic and clinical status information in male subjects affected by HED using a medical questionnaire | Study day 1 - Day of study conduct
Exploratory Objective - To test and refine a computer algorithm for facial recognition of XLHED based on 2D facial photographs | Study day 1 - Day of study conduct
Exploratory Objective - To identify nutritional patterns associated with XLHED | Study day 1 - Day of study conduct
Exploratory Objective - To test for the presence of genetic mutations in a subset of HED-affected subjects enrolled in this study who lack prior genetic diagnosis | Study day 1 - Day of study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy K Grange, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Buenavista Palace Hotel and Spa, Orlando, Florida, United States